CLINICAL TRIAL: NCT02292537
Title: A Phase 3, Randomized, Double-blind, Sham-Procedure Controlled Study to Assess the Clinical Efficacy and Safety of ISIS 396443 Administered Intrathecally in Patients With Later-onset Spinal Muscular Atrophy
Brief Title: A Study to Assess the Efficacy and Safety of Nusinersen (ISIS 396443) in Participants With Later-onset Spinal Muscular Atrophy (SMA)
Acronym: CHERISH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 396443-CS4; 2014-001947-18 (EudraCT Number)
Expanded Access: NCT02865109 (No longer available)
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; SMA; SMN; SMNRx; ISIS-SMNRx; ISIS-SMN Rx; ISIS 396443; CHERISH; IONIS-SMNRx; IONIS-SMN Rx
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nusinersen (Experimental): Nusinersen 12 mg solution via intrathecal (IT) injection on Days 1, 29, 85 and 274.
  Interventions: Drug: Nusinersen
- Sham procedure (Sham Comparator): Sham comparator on Days 1, 29, 85 and 274.
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Drug: Nusinersen — Administered by intrathecal (IT) lumbar puncture (LP) injection
  Other Names: Sprinraza; ISIS 396443; IONIS-SMN Rx; BIIB058
  Arms: Nusinersen
Procedure: Sham procedure — Small needle prick on the lower back at the location where the IT injection is normally made
  Arms: Sham procedure

SUMMARY:
The primary objective of this study is to examine the clinical efficacy of nusinersen (ISIS 396443) administered intrathecally to participants with later-onset Spinal Muscular Atrophy (SMA). The secondary objective is to examine the safety and tolerability of nusinersen administered intrathecally to participants with later-onset SMA.

DETAILED DESCRIPTION:
This study was conducted and the protocol was registered by Ionis Pharmaceuticals, Inc.

In August 2016, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Parent or guardian has signed informed consent and, if indicated per participant's age and institutional guidelines, participant has signed informed assent
* Be medically diagnosed with Spinal Muscular Atrophy (SMA)
* Have onset of clinical signs and symptoms consistent with SMA at greater than 6 months of age
* Be able to sit independently, but has never had the ability to walk independently
* Have Motor Function Score (Hammersmith Functional Motor Scale - Expanded) greater than or equal to 10 and less than or equal to 54 at Screening
* Be able to complete all study procedures, measurements and visits and parent or guardian and subject has adequately supportive psychosocial circumstances, in the opinion of the Investigator
* Have an estimated life expectancy of greater than 2 years from Screening, in the opinion of the Investigator
* Meet age-appropriate institutional criteria for use of anesthesia and sedation, if use is planned for study procedures
* For subjects who have reached reproductive maturity, satisfy study contraceptive requirements

Key Exclusion Criteria:

* Respiratory insufficiency, defined by the medical necessity for invasive or non-invasive ventilation for greater than 6 hours during a 24 hour period, at Screening
* Medical necessity for a gastric feeding tube, where the majority of feeds are given by this route, as assessed by the Site Investigator
* Severe contractures or severe scoliosis evident on X-ray examination at Screening
* Hospitalization for surgery (i.e., scoliosis surgery, other surgery), pulmonary event, or nutritional support within 2 months of Screening or planned during the duration of the study
* Presence of an untreated or inadequately treated active infection requiring systemic antiviral or antimicrobial therapy at any time during the screening period
* History of brain or spinal cord disease, including tumors, or abnormalities by magnetic resonance imaging (MRI) or computed tomography (CT) that would interfere with the LP procedures or cerebrospinal fluid (CSF) circulation
* Presence of an implanted shunt for the drainage of CSF or an implanted central nervous system (CNS) catheter
* History of bacterial meningitis
* Dosing with IONIS-SMN Rx in any previous clinical study
* Prior injury (e.g., upper or lower limb fracture) or surgical procedure which impacts the subject's ability to perform any of the outcome measure testing required in the protocol and from which the subject has not fully recovered or achieved a stable baseline
* Clinically significant abnormalities in hematology or clinical chemistry parameters or electrocardiogram (ECG), as assessed by the Site Investigator, at the Screening visit that would render the subject unsuitable for inclusion
* Treatment with another investigational drug (e.g., oral albuterol or salbutamol, riluzole, carnitine, creatine, sodium phenylbutyrate, et.c), biological agent, or device within 1-month of Screening or 5 half-lives of study agent, whichever is longer. Treatment with valproate or hydroxyurea within 3-months of Screening. Any history of gene therapy, antisense oligonucleotide therapy, or cell transplantation.
* Ongoing medical condition that according to the Site Investigator would interfere with the conduct and assessments of the study. Examples are medical disability (e.g., wasting or cachexia, severe anemia, etc.) that would interfere with the assessment of safety or would compromise the ability of the subject to undergo study procedures.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (24):
- United States (11):
  - UCLA Clinical and Translational Research Center, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Hospital, Orlando, Florida
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia - Neurology, Philadelphia, Pennsylvania
  - Children's Medical Center, Dallas, Texas
- Canada (2):
  - Children's Hospital - London Health Sciences Centre, London, Ontario
  - McGill University Health Centre-Glen Site-CIM, Montreal, Quebec
- Armand Trousseau Hospital, I-Motion, Clinical Trials Platform, Paris, France
- Germany (2):
  - Universitatsklinikum Essen, Essen
  - University Hospital Freiberg, Center for Paediatrics and Adolescent Medicine, Department of Neuropaediatrics and Muscular Disease, Freiburg im Breisgau
- The University of Hong Kong, Queen Mary Hospital, Department of Paediatrics and Adolescent Medicine, Hong Kong, Hong Kong SAR, Hong Kong
- Italy (2):
  - AOU Policlinico G. Martino Dipartimento di Neuroscienze e Centro Clinico Nemo Sud, Messina
  - Fondazione Policlinico Universitario Agostino Gemelli-Universita Cattolica de Sacro Cuore-UOC Neuropsichiatre Infantile, Rome
- Japan (2):
  - Hyogo College of Medicine, Nishinomya-shi, Hyōgo
  - Tokyo Women's Medical University, Shinjuku-ku, Tokyo
- Seoul National University Children's Hospital, Seoul, Korea, South Korea
- Hospital Sant Joan de Deu, Barcelona, Spain
- University of Gothenburg, The Queen Silvia Children's Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Darras BT, Farrar MA, Mercuri E, Finkel RS, Foster R, Hughes SG, Bhan I, Farwell W, Gheuens S. An Integrated Safety Analysis of Infants and Children with Symptomatic Spinal Muscular Atrophy (SMA) Treated with Nusinersen in Seven Clinical Trials. CNS Drugs. 2019 Sep;33(9):919-932. doi: 10.1007/s40263-019-00656-w. PMID 31420846
- [Derived] Mercuri E, Darras BT, Chiriboga CA, Day JW, Campbell C, Connolly AM, Iannaccone ST, Kirschner J, Kuntz NL, Saito K, Shieh PB, Tulinius M, Mazzone ES, Montes J, Bishop KM, Yang Q, Foster R, Gheuens S, Bennett CF, Farwell W, Schneider E, De Vivo DC, Finkel RS; CHERISH Study Group. Nusinersen versus Sham Control in Later-Onset Spinal Muscular Atrophy. N Engl J Med. 2018 Feb 15;378(7):625-635. doi: 10.1056/NEJMoa1710504. PMID 29443664
- See also: Cure SMA — http://www.curesma.org
- See also: Muscular Dystrophy Association — http://mda.org/disease/spinal-muscular-atrophy
- See also: National Organization for Rare Diseases — https://www.rarediseases.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After parental informed consent was obtained and prior to any treatment, participants entered a Screening Period of up to 21 days to determine their eligibility for the study. Of the 179 participants screened, 53 were screening failures.
Period: Overall Study
Arm/Group | Sham Procedure | Nusinersen
Started | 42 | 84
Completed Treatment | 42 | 83 (1 participant completed the study but did not complete treatments due to early study closure)
Completed | 42 | 84
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Set: All participants who were randomized and received at least 1 dose of study drug/sham procedure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Procedure | Nusinersen | Total
Number analyzed (Participants) | 42 | 84 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.4 (1.61) | 3.8 (1.63) | 3.6 (1.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 46 | 67
  Male | 21 | 38 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 42 | 80 | 122
  Asian | 7 | 16 | 23
  Black | 1 | 1 | 2
  White | 30 | 64 | 94
  Multiple | 4 | 3 | 7
Hammersmith Functional Motor Scale - Expanded (HFMSE) Score [Mean (Standard Deviation); unit: scores on a scale] — The HFMSE consists of 33 scored activities used to assess motor function in children with SMA. Participants were asked to do a specific activity (such as rolling) and they were then graded on the quality and execution of that movement on a scale of 0=being unable, 1=performed with some compensation, and 2=unaided. The overall score is the sum of the scores for all activities with a maximum achievable score of 66. Higher scores indicate increased motor function.
  scores on a scale | 19.9 (7.23) | 22.4 (8.33) | 21.6 (8.03)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hammersmith Functional Motor Scale - Expanded (HFMSE) Score at Month 15
Description: The HFMSE consists of 33 scored activities used to assess motor function in children with SMA. The scale was originally developed with 20 scored activities and was devised for use in children with SMA Type 2 and Type 3 with limited ambulation to give objective information on motor ability and clinical progression. The expanded scale includes an additional module of 13 items developed to allow for evaluation of ambulatory SMA patients. Participants were asked to do a specific activity (such as rolling) and they were then graded on the quality and execution of that movement on a scale of 0=being unable, 1=performed with some compensation, and 2=unaided. The overall score is the sum of the scores for all activities with a maximum achievable score of 66. Higher scores indicate increased motor function. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Month 15
Population: ITT Set: All participants who were randomized and received at least 1 dose of study drug/sham procedure. Missing postbaseline HFMSE data were imputed using the multiple imputation method.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sham Procedure | Nusinersen
Number analyzed (Participants) | 42 | 84
scores on a scale | -1.0 [-2.5 to 0.5] | 3.9 [3.0 to 4.9]
Statistical Analysis 1: Comparison: Sham Procedure vs Nusinersen; Test type: Superiority; p = 0.0000001, ANCOVA; ANCOVA model with treatment group as a factor and age at Screening and baseline HFMSE score as covariates; LS Mean Difference = 4.9, 95% CI 2-sided [3.1 to 6.7], Standard Error of Mean 0.91

2. Secondary Outcome: Proportion of Participants Who Achieved a 3-Point Increase From Baseline in HFMSE Score at Month 15
Description: as for outcome 1
Time Frame: Baseline and Month 15
Population: ITT Set: All participants who were randomized and received at least 1 dose of study drug/sham procedure. Missing postbaseline HFMSE data were imputed using multiple imputation.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Sham Procedure | Nusinersen
Number analyzed (Participants) | 42 | 84
Proportion of participants | 26.3 [12.40 to 40.22] | 56.8 [45.62 to 68.05]
Statistical Analysis 1: Comparison: Sham Procedure vs Nusinersen; Test type: Superiority; p = 0.0006, Regression, Logistic — Based on multiple imputation and logistic regression with treatment effect and adjustment for each participant's age at screening and HFMSE score at baseline; Odds Ratio (OR) = 5.59, 95% CI 2-sided [2.09 to 14.91]
Statistical Analysis 2: Comparison: Sham Procedure vs Nusinersen; Test type: Superiority; Difference in Proportions = 30.5, 95% CI 2-sided [12.74 to 48.31] — Difference in proportions of Nusinersen minus Sham Procedure are from multiple imputation procedure and are based on binomial proportions

3. Secondary Outcome: Proportion of Participants That Achieved Any New Motor Milestone at Month 15
Description: New motor milestones are defined as sitting without support, hands-and-knees crawling, standing with assistance, walking with assistance, standing alone and walking alone.
Time Frame: Month 15
Population: Efficacy Set: All participants with a Day 456 Visit and all participants with a time difference of at least 463 days (456 days plus a 7-day window) between the date of first dose and the date for the final analysis. Based on imputed data where there was missing data.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Sham Procedure | Nusinersen
Number analyzed (Participants) | 34 | 66
Proportion of participants | 5.9 [0.72 to 19.68] | 19.7 [10.93 to 31.32]
Statistical Analysis 1: Comparison: Sham Procedure vs Nusinersen; Test type: Superiority; p = 0.0811, Fisher Exact; Difference in Proportions = 13.8, 95% CI 2-sided [-6.64 to 34.17] — Difference in proportions of Nusinersen minus Sham Procedure is based on exact unconditional confidence interval

4. Secondary Outcome: Number of New Motor Milestones Achieved Per Participant
Description: as for outcome 3
Time Frame: Month 15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milestones achieved
Arm/Group | Sham Procedure | Nusinersen
Number analyzed (Participants) | 34 | 66
milestones achieved | -0.2 (0.54) | 0.2 (0.51)
Statistical Analysis 1: Comparison: Sham Procedure vs Nusinersen; Test type: Superiority; LS Mean Difference = 0.4, 95% CI 2-sided [0.2 to 0.7] — Based on ANCOVA with treatment as a fixed effect and adjustment for each participant's age at screening and number of milestones at baseline

5. Secondary Outcome: Change From Baseline in Revised Upper Limb Module (RULM) Test
Description: The RULM Test is used in patients with SMA to assess upper limb functional ability items that are reflective of activities of daily living (i.e., raise a can to mouth as if drinking, take a coin and place it in a box, remove the lid of a container). The RULM test has a total of 20 items with an entry item that serves as functional class identification and does not contribute to the total score. The remaining 19 scorable items reflect different functional domains and are graded on a 3-point system with a score of 0 (unable), 1 (able, with modification), and a maximum of 2 (able, no difficulty). There is only 1 item (item I) that is scored as a can/cannot score, with 1 as the highest score. Scorable items are summed for a total score range of 0-37, with higher scores increased great upper limb function. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Month 15
Population: ITT Set: All participants who were randomized and received at least 1 dose of study drug/sham procedure. Missing postbaseline data were imputed using multiple imputation.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sham Procedure | Nusinersen
Number analyzed (Participants) | 42 | 84
scores on a scale | 0.5 [-0.6 to 1.6] | 4.2 [3.4 to 5.0]
Statistical Analysis 1: Comparison: Sham Procedure vs Nusinersen; Test type: Superiority; LS Mean Differenec = 3.7, 95% CI 2-sided [2.3 to 5.0] — From multiple imputation procedure, based on ANCOVA with treatment as a fixed effect and adjustment for each participant's age at screening and derived total score at baseline

6. Secondary Outcome: Proportion of Participants That Achieved Standing Alone
Description: If the participant was unable to achieve standing alone at Baseline but could achieve this at Month 15 then they were considered a responder. If they could not achieve this or if a participant terminated the study prior to the 15-month assessment due to treatment failure or death, then any imputed value was ignored and the participant was considered as a non-responder.
Time Frame: Month 15
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Sham Procedure | Nusinersen
Number analyzed (Participants) | 34 | 66
Proportion of participants | 2.9 [0.07 to 15.33] | 1.5 [0.04 to 8.16]
Statistical Analysis 1: Comparison: Sham Procedure vs Nusinersen; Test type: Superiority; Difference in Proportions = -1.4, 95% CI 2-sided [-21.84 to 19.34] — Difference in proportions of Nusinersen minus Sham Procedure is based on exact unconditional confidence interval

7. Secondary Outcome: Proportion of Participants That Achieved Walking With Assistance
Description: If the participant was unable to achieve walking with assistance at baseline but could achieve this at Month 15 then they were considered a responder. If they could not achieve this or if a participant terminated the study prior to the 15-month assessment due to treatment failure or death, then any imputed value was ignored and the participant was considered as a non-responder.
Time Frame: Month 15
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Sham Procedure | Nusinersen
Number analyzed (Participants) | 34 | 66
Proportion of participants | 0.0 [0.00 to 10.28] | 1.5 [0.04 to 8.16]
Statistical Analysis 1: Comparison: Sham Procedure vs Nusinersen; Test type: Superiority; Difference in Proportions = 1.5, 95% CI 2-sided [-19.10 to 22.10] — Difference in proportions of Nusinersen minus Sham Procedure is based on exact unconditional confidence interval

8. Secondary Outcome: Number of Participants That Experienced Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AEs: any sign, symptom, or diagnosis/disease that is unfavorable or unintended, that is new, or if pre-existing, worsens in participants administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. SAEs: an event that results in death; an event that, in the view of the investigator, places the participant at immediate risk of death; an outcome that results in a congenital anomaly/birth defect diagnosed in a child of a participant; an event that requires or prolongs inpatient hospitalization; an event that results in persistent or significant disability/incapacity. Any other medically important event that, in the opinion of the investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above.
Time Frame: Baseline through Month 15
Population: Safety Set: All participants who were randomized and received at least 1 dose of study drug/sham procedure. All participants with AEs were reported in this outcome measure, whereas in Adverse Event section there was at 5% reporting threshold to be met.
Measure: Number; unit: participants
Arm/Group | Sham Procedure | Nusinersen
Number analyzed (Participants) | 42 | 84
participants
  AEs | 42 | 78
  SAEs | 12 | 14

9. Secondary Outcome: Number of Participants With Clinically Significant Vital Sign Abnormalities
Description: Vital signs assessed for clinical significance include resting blood pressure, pulse, respiratory rate, and temperature.
Time Frame: Baseline through Month 15
Population: Safety Set: All participants who were randomized and received at least 1 dose of study drug/sham procedure. Any new or worsening vital sign findings were reported as AEs and are presented in the AE/SAE section of the results.
Measure: Number; unit: participants
Arm/Group | Sham Procedure | Nusinersen
Number analyzed (Participants) | 42 | 84
participants
  Systolic blood pressure <90 mmHg | 33 | 80
  Systolic blood pressure >140 mmHg | 1 | 4
  Systolic blood pressure >160 mmHg | 0 | 2
  Diastolic blood pressure <50 mmHg | 31 | 65
  Diastolic blood pressure >90 mmHg | 7 | 11
  Diastolic blood pressure >100 mmHg | 2 | 2
  Heart rate <60 beats/min | 0 | 1
  Heart rate >100 beats/min | 42 | 84
  Temperature >38.0 C | 4 | 10
  Temperature <36.0 C | 14 | 33
  Respiratory rate <12 breaths/min | 0 | 1
  Respiratory rate >20 breaths/min | 42 | 84

10. Secondary Outcome: Number of Participants With Clinically Significant Weight Abnormalities
Description: Weight changes assessed from Baseline to Month 15.
Time Frame: Baseline through Month 15
Population: Safety Set: All participants who were randomized and received at least 1 dose of study drug/sham procedure. Any new or worsening weight abnormality findings were reported as AEs and are presented in the AE/SAE section of the results.
Measure: Number; unit: participants
Arm/Group | Sham Procedure | Nusinersen
Number analyzed (Participants) | 42 | 84
participants
  Weight decrease of >=7% from baseline | 3 | 4
  Weight increase of >=7% from baseline | 38 | 77

11. Secondary Outcome: Number of Participants With Clinically Significant Neurological Examination Abnormalities
Description: Neurological changes assessed for clinical significance include assessment of mental status, level of consciousness, sensory function, motor function, cranial nerve function, and reflexes.
Time Frame: Baseline through Month 15
Population: Safety Set: All participants who were randomized and received at least 1 dose of study drug/sham procedure. Neurological examination clinical significance was not collected.
Arm/Group | Sham Procedure | Nusinersen
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Abnormalities
Description: Physical examination changes were assessed for clinical significance.
Time Frame: Baseline through Month 15
Population: Safety Set: All participants who were randomized and received at least 1 dose of study drug/sham procedure. Physical examination clinical significance was not collected.
Arm/Group | Sham Procedure | Nusinersen
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Parameter Abnormalities
Description: Laboratory parameter changes assessed for clinical significance include serum chemistry, hematology, coagulation and urinalysis.
Time Frame: Baseline through Month 15
Population: Safety Set: All participants who were randomized and received at least 1 dose of study drug/sham procedure. Any new or worsening clinical laboratory parameter findings were reported as AEs and are presented in the AE/SAE section of the results.
Measure: Number; unit: participants
Arm/Group | Sham Procedure | Nusinersen
Number analyzed (Participants) | 42 | 84
participants
  Hematology: Hemoglobin - High | 2 | 2
  Hematology: Hemoglobin - Low | 7 | 15
  Hematology: Hematocrit - High | 3 | 1
  Hematology: Hematocrit - Low | 6 | 18
  Hematology: Red blood cells - High | 2 | 2
  Hematology: Red blood cells - Low | 7 | 13
  Hematology: White blood cells - High | 11 | 12
  Hematology: White blood cells - Low | 10 | 20
  Hematology: Platelet Count - High | 5 | 10
  Hematology: Platelet count - Low | 10 | 15
  Blood Chemistry: Bilirubin - Low | 19 | 36
  Blood Chemistry: Bilirubin - High | 1 | 0
  Blood Chemistry: Total bilirubin - direct - Low | 5 | 8
  Blood Chemistry: Total bilirubin - direct - High | 0 | 0
  Blood Chemistry: Total bilirubin - indirect- Low | 0 | 0
  Blood Chemistry: Total bilirubin - indirect- High | 1 | 0
  Blood Chemistry: Alkaline phosphatase - Low | 1 | 10
  Blood Chemistry: Alkaline phosphatase - High | 0 | 0
  Blood Chemistry: ALT - Low | 0 | 1
  Blood Chemistry: ALT - High | 4 | 3
  Blood Chemistry: AST - Low | 0 | 0
  Blood Chemistry: AST- High | 2 | 3
  Blood Chemistry: BUN - Low | 0 | 2
  Blood Chemistry: BUN - High | 1 | 2
  Blood Chemistry: Creatinine - Low | 17 | 39
  Blood Chemistry: Creatinine- High | 0 | 1
  Blood Chemistry: Sodium - Low | 1 | 1
  Blood Chemistry: Sodium - High | 0 | 0
  Blood Chemistry: Potassium - Low | 2 | 0
  Blood Chemistry: Potassium - High | 1 | 0
  Blood Chemistry: Chloride - Low | 0 | 0
  Blood Chemistry: Chloride - High | 0 | 0
  Blood Chemistry: Total protein - Low | 1 | 7
  Blood Chemistry: Total protein - High | 9 | 13
  Blood Chemistry: Albumin - Low | 0 | 0
  Blood Chemistry: Albumin - High | 19 | 27
  Blood Chemistry: Calcium - Low | 0 | 1
  Blood Chemistry: Calcium - High | 9 | 20
  Blood Chemistry: Phosphorus - Low | 0 | 0
  Blood Chemistry: Phosphorus - High | 8 | 8
  Blood Chemistry: Bicarbonate - Low | 11 | 29
  Blood Chemistry: Bicarbonate - High | 0 | 0
  Blood Chemistry: Glucose - Low | 7 | 17
  Blood Chemistry: Glucose - High | 26 | 44
  Blood Chemistry: Cystatin C - Low | 18 | 36
  Blood Chemistry: Cystatin C -High | 0 | 1
  Blood Chemistry: CPK - Low | 0 | 0
  Blood Chemistry: CPK - High | 10 | 16
  Urinalysis: Specific gravity - Low | 0 | 0
  Urinalysis: Specific gravity - High | 2 | 1
  Urinalysis: pH- Low | 0 | 0
  Urinalysis: pH - High | 0 | 0
  Urinalysis: Protein - High | 14 | 43
  Urinalysis: Glucose - High | 2 | 2
  Urinalysis: Ketones - High | 18 | 29
  Urinalysis: Bilirubin - High | 0 | 0
  Urinalysis: Blood - High | 1 | 1
  Urinalysis: RBC - High | 1 | 6
  Urinalysis: WBC - High | 4 | 13
  Urinalysis: Epithelial Cells - High | 0 | 0
  Urinalysis: Bacteria - High | 15 | 24
  Urinalysis: Casts - High | 0 | 0
  Urinalysis: Hyaline casts - High | 1 | 5
  Urinalysis: Crystals - High | 0 | 0
  Urinalysis: Amorphous crystals - High | 10 | 16
  Urinalysis: Calcium oxalate crystals - High | 17 | 26
  Urinalysis: Uric acid crystals - High | 5 | 5

14. Secondary Outcome: Number of Participants With Abnormal, Clinically Relevant Post-Baseline Worsening in Electrocardiogram (ECG) in Results
Description: The number of participants with abnormal, clinically relevant worsening, defined as participants with an ECG interpreted as abnormal and clinically relevant, with a comparison with Baseline value is reported.
Time Frame: Baseline through Month 15
Population: Safety Set: All participants who were randomized and received at least 1 dose of study drug/sham procedure.
Measure: Number; unit: participants
Arm/Group | Sham Procedure | Nusinersen
Number analyzed (Participants) | 42 | 84
participants | 2 | 0

15. Secondary Outcome: Number of Participants Taking Any Concomitant Medication Related to Dosing Procedure or Sham Procedure
Description: Concomitant medications include prescription and over-the-counter medications administered to participants on or after the first day of study treatment.
Time Frame: Baseline through Month 15
Population: Safety Set: All participants who were randomized and received at least 1 dose of study drug/sham procedure.
Measure: Number; unit: participants
Arm/Group | Sham Procedure | Nusinersen
Number analyzed (Participants) | 42 | 84
participants | 42 | 84

ADVERSE EVENTS:
Time Frame: From signing of Informed Consent to the end of the Follow-up period (Month 15)
Description: Treatment emergent AEs are presented regardless of seriousness or relationship to investigational product.
Arm/Group | Sham Procedure | Nusinersen
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/84
Serious Adverse Events (participants affected / at risk) | 12/42 | 14/84
Other Adverse Events (participants affected / at risk) | 42/42 | 75/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Procedure (N=42) | Nusinersen (N=84)
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 2 | 0
Pain (General disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 2 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 2
Pneumonia adenoviral (Infections and infestations) | 1 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 3
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Procedure (N=42) | Nusinersen (N=84)
Constipation (Gastrointestinal disorders) | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 8
Vomiting (Gastrointestinal disorders) | 5 | 24
Pyrexia (General disorders) | 15 | 36
Bronchitis (Infections and infestations) | 4 | 7
Conjunctivitis (Infections and infestations) | 2 | 6
Ear infection (Infections and infestations) | 5 | 7
Gastroenteritis (Infections and infestations) | 8 | 9
Gastroenteritis viral (Infections and infestations) | 4 | 8
Influenza (Infections and infestations) | 2 | 8
Nasopharyngitis (Infections and infestations) | 15 | 20
Otitis media (Infections and infestations) | 4 | 5
Pharyngitis streptococcal (Infections and infestations) | 3 | 4
Pneumonia (Infections and infestations) | 6 | 4
Upper respiratory tract infection (Infections and infestations) | 19 | 25
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 21
Joint contracture (Musculoskeletal and connective tissue disorders) | 7 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4
Scoliosis (Musculoskeletal and connective tissue disorders) | 3 | 3
Headache (Nervous system disorders) | 3 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 5

LIMITATIONS AND CAVEATS:
After the interim analysis of the study, the decision was made in October 2016 to terminate the study early and participants were invited for end-of-study visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT02292537/SAP_000.pdf
  • Study Protocol (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT02292537/Prot_001.pdf